CLINICAL TRIAL: NCT05422209
Title: The Influence of Simultaneous Posterior Colporrhaphy and Perineoplasty on the Efficiency and Safety of Mesh-augmented Sacrospinal Fixation (Apical Sling) in Advanced POP Repair. Randomized Controlled Study.
Brief Title: The Influence of Simultaneous Posterior Colporrhaphy and Perineoplasty on the Efficiency and Safety of Mesh-augmented Sacrospinal Fixation (Apical Sling) in Advanced POP Repair.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Shkarupa Dmitry, Ph.D., Deputy Director for medical care, Chief Urologist of Saint Petersburg State University Clinic of advanced medical technologies n.a. N.I.Pirogov., Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSF and perineoplasty
Record Dates: First submitted 2022-05-18; First posted 2022-06-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; vaginal repair; vaginal mesh; sacrospinous fixation; colporrhaphy; perineoplasty
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesh-augmented sacrospinal fixation with posterior colporrhaphy and perineoplasty. (Active Comparator)
  Interventions: Procedure: Mesh-augmented sacrospinal fixation with posterior colporrhaphy and perineoplasty.
- Mesh-augmented sacrospinal fixation with posterior colporrhaphy. (Active Comparator)
  Interventions: Procedure: Mesh-augmented sacrospinal fixation with posterior colporrhaphy.

INTERVENTIONS:
Procedure: Mesh-augmented sacrospinal fixation with posterior colporrhaphy and perineoplasty. — Vaginal mesh-augmented sacrospinal fixation with posterior colporrhaphy and perineoplasty.
  Arms: Mesh-augmented sacrospinal fixation with posterior colporrhaphy and perineoplasty.
Procedure: Mesh-augmented sacrospinal fixation with posterior colporrhaphy. — Vaginal mesh-augmented sacrospinal fixation with posterior colporrhaphy.
  Arms: Mesh-augmented sacrospinal fixation with posterior colporrhaphy.

SUMMARY:
This is a prospective randomized controlled study, designed to assess the influence of posterior colporrhaphy and perineoplasty performed simultaneously with mesh-augmented sacrospinal fixation (apical sling) in advanced pelvic organ prolapse repair.

DETAILED DESCRIPTION:
BACKGROUND Pelvic organ prolapse (POP) is revealed by the gynecological examination in 40-60 % of parous women. A pelvic floor defect is represented by cystocele almost in a half of cases. At the same time it is known that just the loss of apical support favors going out of the anterior vaginal wall beyond the hymen. Today the vast majority of specialists share one view that the uterus with its sacral-uterine-cardinal ligament complex is a key element for the reliable support of the pelvic floor. It is also considered that perineal body insufficiency promotes the development of POP because the small pelvic organs do not have support on which they could lie. The perineal body is a part of the support level III according to DeLancey. Hiatus enlargement is associated with damage of the elevator muscle of anus and one of the factors for POP development both at a clinical examination and ultrasound scanning. Perineoplasty is one of the methods for correction of hiatus opening and anatomical perineal body insufficiency. An important aspect in POP surgery consists in prevention of a recurrence after the surgical treatment. It is important to mention that today there are no randomized studies comparing the efficiency of transvaginal pelvic floor reconstruction using a mesh for apical fixation with and without the recovery of the support level 3 according to DeLancey. Thus, understanding of mechanisms for prevention of repeated surgeries is fundamental and essential for successful treatment of POP.

PREOPERATIVE ASSESSMENT All patients who meet eligibility criteria will undergo a preoperative assessment: medical history, physical and vaginal examination, assessing pelvic organ prolapse according to Pelvic Organ Prolapse Quantification System (POP-Q). All patients will complete questionnaires validated in Russia: Pelvic Floor Disability Index (PFDI-20), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, short form (PISQ-SF), Patient Global Impression of Improvement (PGI-I).

MATERIALS AND METHODS Our hypothesis is that posterior colporrhaphy and perineoplasty performed simultaneously with mesh-augmented sacrospinal fixation reduces POP recurrence in any compartment.

Taking into account the available data on frequency of recurrences after unilateral sacrospinal fixation according to hybrid technology (7.4 %) and also clinical observation on frequency of recurrences after three-level hybrid reconstruction (1 %), study power of 80 %, significance level of 5 %, 282 patients are necessary to confirm an expected difference in frequency of recurrences. In order to compensate data losses, the calculated sample size was increased by 10 %. As a result, the total sample size is 310 patients.

All enrolled patients will be randomly assigned to mesh-augmented sacrospinal fixation with posterior colporrhaphy or sacrospinal fixation with posterior colporrhaphy and perineoplasty treatment groups in equal ratio the day before the surgery, using computer randomization.

All data will be collected by medical staff not involved in treatment. Collected pre- and postoperative data will be anonymized using unique codes, that patients will receive immediately after randomization.

All surgical interventions will be performed by 4 qualified surgeons. Postoperative follow-up will be performed 6, 12 and 24 months after surgery by 2 researchers, who will be blinded about the type of intervention.

ELIGIBILITY:
Inclusion Criteria:

* The age of a subject is 45 to 80 years.
* Leading point of prolapse is at the level of the hymen or distal to the hymen (Ba, C>=0 according to POP-Q classification)
* Patient's ability to read and sign the informed consent form.
* Socialized patient who is able to fill in validated questionnaires and arrive for control postoperative examination in future.
* Patient's consent for participation in the study.

Exclusion Criteria:

* The subject has presence of oncologic disease which was diagnosed earlier or is active now.
* The subject had prior surgery for POP, SUI or hysterectomy
* The subject has gynecological deseases (recurrent uterine bleeding, endometrial hyperplasia, the presence of atypical cells in cervical smears, adenomyosis, multiple uterine myoma)
* The subject has urinary incontinence
* The subject is planning pregnancy
* The subject has an active urinary tract infection or skin infection in the region of surgery or acute infectious desease
* The subject is unable to visit postoperative check-ups
* Refusal from participation.
* Bp > C according to POP-Q system.
* gh < 4 cm and > 6 cm according to POP-Q system.

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-03-09 (Actual); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
Objective cure rate | 24 months (2 years)
  The patient is considered cured if there is no prolapse beyond the hymen and the cervix is above -1 cm according to POP-Q (0-1 stage)

SECONDARY OUTCOMES:
Satisfaction with the surgery | Measured postoperatively at intervals of 6, 12 and 24 months postoperatively
  Measured through the Patient Global Impression of Improvement questionnaire (PGI-I), validated in Russia. The patient marks the number that best describes her post-operative condition, compared with how it was before surgery. The score ranges from 1 (very much better) to 7 (very much worse).
The impact of treatment on sexual function | Measured postoperatively at intervals of 6, 12 and 24 months postoperatively
  Measured through the scoring of Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) validated in Russia. The scale evaluates sexual function in patients with urinary incontinence and/or POP. The responses are graded on a five-point Likert scale ranging from 0 (always) to 4 (never). Items 1 - 4 are reversely scored and a total of 48 is the maximum score. The higher scores indicate better sexual function.
The impact of treatment on the quality of life | Measured postoperatively at intervals of 6, 12 and 24 months postoperatively
  Measured through the Pelvic Floor Disability Index (PFDI-20), validated in Russia. The item includes 20 questions. The score ranges from 0 to 300. The higher the score, the worse the outcome.
Observed complications | Measured postoperatively at intervals of 6, 12 and 24 months postoperatively
  Presence of any adverse effects such as: bleeding requiring blood transfusion, haematoma, organ perforation, nerve injury, vaginal scarring and shortening, wound infection, urinary tract infection, pelvic pain, mesh extrusion in the vagina, mesh erosion into the urinary tract, dyspareunia de novo, de novo urgency, atonic bladder, de novo stress urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Shkarupa, MD, PhD, Study Chair — Saint Petersburg State University, Russia
Locations (1):
- Saint-Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shakhaliev RA, Shulgin AS, Kubin ND, Kondratiev AS, Suchkov DA, Neklasova SV, Shkarupa DD. The influence of simultaneous posterior colporrhaphy and perineoplasty on the efficiency and safety of mesh-augmented sacrospinal fixation (apical sling) in advanced POP repair. Trials. 2024 Oct 2;25(1):647. doi: 10.1186/s13063-024-08448-4. PMID 39358750